CLINICAL TRIAL: NCT04417595
Title: Investigating N-3 Fatty Acids to Prevent Neonatal Tobacco-related outcomeS
Brief Title: Omega-3 Fatty Acids for Smoking Cessation in Pregnancy
Acronym: INFANTS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Harvey Murff, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200609; R01HD098719 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Preterm Labor; Tobacco Use Disorder
MeSH Terms: conditions — Obstetric Labor, Premature; Tobacco Use Disorder | interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomizes, parallel arm, double-blind, placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish Oil (Experimental): Participants allocated to n-3 LCPUFA supplementation will be instructed to take four 1000 mg n-3 LCPUFA capsules (Metagenics™) daily. This will provide a total daily dose of 4000 mg n-3 LCPUFAs (2840 EPA and 1160 DHA).
  Interventions: Drug: Fish Oil (Containing Omega-3 Acids)
- Olive Oil (Placebo Comparator): Oleic acid (olive oil) capsules have a similar texture, size, color, and consistency to EPA capsules. Participant will be instructed to take four 100mg olive oil capsules
  Interventions: Drug: Olive Oil

INTERVENTIONS:
Drug: Fish Oil (Containing Omega-3 Acids) — Fish Oil Supplement
  Other Names: Fish Oil
  Arms: Fish Oil
Drug: Olive Oil — Olive Oil Supplement
  Other Names: Placebo
  Arms: Olive Oil

SUMMARY:
Smoking is the most important modifiable risk factor for adverse pregnancy outcomes including preterm birth, neonatal death, and maternal complications. Rates of smoking cessation during pregnancy are low, particularly in underserved populations, and currently approved pharmacotherapies for smoking cessation either are considered unsafe in pregnancy or have uncertain effectiveness. Identifying safe and effective interventions, which might mitigate the adverse effects of smoking on maternal-fetal outcomes, is a major public health priority. We hypothesize that smoking-induced n-3 LCPUFA relative deficiencies may be an important mechanism contributing to tobacco-related adverse pregnancy outcomes and that n-3 LCPUFA supplementation specifically targeted to pregnant smokers may reduce these complications. Support for this hypothesis comes from a recent secondary analysis of the Omega-3 Fatty Acids Supplementation to Prevent Preterm Birth trial that found that only smokers taking n-3 LCPUFAs had a reduction in preterm labor risk as compared to non-smokers. While compelling, this study was a post hoc analysis that included only a small sample of smokers and did not collect data on smoking behaviors during follow up. Yet the ascertainment of longitudinal smoking behavior is critical, as some clinical studies have found that supplemental n-3 LCPUFAs might also reduce nicotine cravings, and lower daily cigarette use. Thus, smokers may doubly benefit from replenishing n-3 LCPUFAs via lower risk of preterm labor and/or increased smoking cessation. To address these knowledge gaps, we are proposing a multi-center, randomized, placebo-controlled, double-blinded study of n-3 LCPUFA supplementation in 400 pregnant smokers. We will collect detailed information on smoking behavior, validated biological markers of cigarette exposure (urinary cotinine, end-expiratory carbon monoxide) and biomarkers of n-3 LCPUFA status (red blood cell phospholipid membrane fatty acids). Our specific aims of this proposal are to 1) determine the effect of supplemental n-3 LCPUFAs on gestational age at delivery and preterm labor in pregnant smokers and 2) determine the effect of n-3 LCPUFA supplementation on tobacco use in pregnant smokers. We will recruit potential participants from eight obstetrics clinics across the Middle-Tennessee area. Our study could have a major translational impact on both adverse tobacco-related birth outcomes and smoking cessation efforts.

DETAILED DESCRIPTION:
Tobacco use is the most important modifiable risk factor associated with adverse pregnancy outcomes and increases the risk of preterm birth, intrauterine growth restriction and sudden infant death syndrome. Over 11% of women report smoking during pregnancy, with higher rates seen in the Southeastern United States. Fewer than half of pregnant smokers are able to quit on their own during pregnancy. Currently, FDA-approved pharmacological strategies for smoking cessation are generally not used in pregnancy: varenicline and bupropion are unsafe and nicotine replacement therapy has limited data to support its efficacy in pregnant smokers. Identifying safe and effective therapies to prevent tobacco-related pregnancy outcomes and/or increase smoking cessation in pregnant women would have a substantial public health impact.

Our group and others have reported that cigarette smoking is associated with a relative deficiency in circulating n-3 long-chain polyunsaturated fatty acid (n-3 LCPUFA) levels. Our overarching hypothesis is that smoking-induced n-3 LCPUFA deficiencies contribute to tobacco-related adverse pregnancy outcomes and that supplementation of n-3 LCPUFAs in pregnant smokers may prevent these complications. Support for this hypothesis comes from a recent secondary analysis of the Omega-3 Fatty Acids Supplementation to Prevent Preterm Birth trial which found that only smokers taking n-3 LCPUFAs had a reduction in preterm labor risk as compared to non-smokers. While compelling, this study was a post hoc analysis that included only a small sample of smokers and did not collect data on smoking behaviors during follow up. Yet the ascertainment of longitudinal smoking behavior is critical, as some clinical studies have found that supplemental n-3 LCPUFAs might also reduce nicotine cravings and lower daily cigarette use. Thus, smokers may doubly benefit from replenishing n-3 LCPUFAs via lower risk of preterm labor and/or increased smoking cessation. We conducted a placebo-controlled pilot RCT of n-3 LCPUFAs in 28 pregnant smokers and found the intervention to be feasible and well-tolerated. Compared to placebo, n-3 LCPUFAs lowered both nicotine dependence at 4 weeks (change from baseline in Fagerström Test for Nicotine Dependence -2.5 vs. 0, p = 0.01) and resulted in a non-statistically significant reduction in cigarettes per day and urine cotinine. To address important remaining knowledge gaps we propose the Investigating N-3 Fatty Acids to prevent Neonatal Tobacco related outcomeS (INFANTS).

Our proposal has three Specific Aims.

Specific Aim 1: To determine the effect of supplemental n-3 LCPUFAs compared to placebo on gestational age at delivery and preterm labor in pregnant smokers.

Specific Aim 2: To determine the effect of supplemental n-3 LCPUFAs compared to placebo on tobacco use in pregnant smokers.

Specific Aim 3: To determine if the effect of supplemental n-3 LCPUFAs on preterm labor is mediated by changes in smoking behavior and/or increases in circulating n-3 LCPUFAs.

The INFANTS study is a multicenter, randomized, double-blind, placebo controlled study that will randomize 400 pregnant smokers to either supplemental n-3 LCPUFAs or placebo. Participants will be enrolled between 12 and 24 weeks gestation and followed until delivery. We will recruit participants from eight clinical centers in the Middle-Tennessee area. We will assess smoking behavior after 12-weeks of supplementation using self-report and validated biomarkers of tobacco exposure (urine cotinine). We will measure response to supplementation using biological markers of n-3 LCPUFA status (red blood cell phospholipid membrane fatty acid percentages). Our primary endpoint will be preterm labor as reflected by gestational age at delivery, which will be extracted from the medical record. Our secondary endpoint will be change from baseline in cigarettes per day at 12 weeks biochemically confirmed through reduction in urine cotinine. We will conduct mediation analysis to better understand the mechanisms contributing to the effects of supplemental n-3 LCPUFAs on birth outcomes in pregnant smokers.

Our study is innovative in that it will be the first clinical trial of n-3 LCPUFAs exclusively recruiting pregnant smokers. This will be the first study to evaluate the impact on n-3 LCPUFAs on tobacco use in smokers who wish to quit, thus identifying a novel strategy to reduce tobacco use that could be relevant for all smokers.

n-3 LCPUFAs supplements are well tolerated in pregnancy but currently are not recommended as part of routine prenatal care in smokers. Thus if our study demonstrated that supplemental n-3 LCPUFAs are effective at reducing the risk of tobacco-related adverse neonatal outcomes and/or reducing tobacco use during pregnancy, our results could have an immediate and major clinical impact on pregnancy care and neonatal outcomes in the United States.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 or ≤ 40 years of age
* Currently reporting daily cigarette use (≥ 1 CPD; reporting 10 or more CPD prior to pregnancy)
* Between 12 and 24 weeks gestation
* An exhaled carbon monoxide reading of at least 8 ppm
* A cell phone or land line that can be reached directly

Exclusion Criteria:

* Allergy to fish; currently using fish oil supplements
* Active substance abuse (not including supervised buprenorphine use)
* Unable to give consent or obtain assent for minors
* Known fetal abnormality
* Chronic hypertension
* Seizure disorder
* Clotting disorder
* White's classification D or higher diabetes
* Planned cerclage
* Plan move from the Middle-Tennessee area within the next 9-months
* Insufficient time to perform the complete enrollment process
* Barrier to communication (e.g., low English proficiency or hearing/speech impairment)

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Actively pregnant
Enrollment: 400 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery | At delivery
  Gestational age at randomization will be determined on the basis of the last menstrual period and earliest ultrasound examination and will not be revised after being assigned a study group. Gestational age will be estimated from the last menstrual period (LMP) and adjusted for the first-trimester ultrasound. If a self-reported LMP is greater than 7 days from the calculated ultrasound LMP, the ultrasound will be used to assign gestational age.
Change in cigarettes per day | At 12 weeks
  Percentage change from baseline in cigarettes per day (CPD) at 12 weeks. The outcome will be determined based on participant self-report.

SECONDARY OUTCOMES:
Percent of neonates with fetal death and still birth | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Individualized birth weight Z-score (adjusted for gestational age and maternal weight) | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. Birth weight will be collected in kilograms. Maternal weight will be collected in kilograms and obtained from medical record review.
Apgar score | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (Score ranges from 0 to 10).
Percent of neonates with intraventricular hemorrhage | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of neonates with neonatal enterocolitis | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of neonates with a congenital abnormality | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of neonates with neonatal respiratory distress | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of participants with maternal mortality | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of participants requiring cesarean delivery | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of participants developing hypertension in pregnancy | At delivery
  Obtained from medical record review of delivery records by study personnel blinded to treatment allocation. This will be a categorical variable (yes or no). Outcomes will be adjudicated by study obstetricians blinded to treatment allocation.
Percent of participants reaching point prevalence abstinence | At 12 weeks
  Point prevalence abstinence at 12 weeks will be based on self-reported smoking cessation and biochemically confirmed by end-expired carbon monoxide ( end-expired CO less than 4 ppm
Percent of patients with a decrease in self-reported nicotine dependence | At 12 weeks
  Changes in nicotine dependence based on changes in the Fagerström Test for Nicotine Dependence.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murff HJ, Greevy RA, Sanghani RS, Hartmann KE, Hartert TV, Graves CR, Lee SS, Tindle HA. Investigating N-3 Fatty Acids to prevent Neonatal Tobacco-related outcomeS (INFANTS): study protocol for a double-blind, randomized, placebo-controlled parallel clinical trial of n-3 polyunsaturated fatty acids in pregnant smokers. Trials. 2021 Dec 14;22(1):922. doi: 10.1186/s13063-021-05865-7. PMID 34906201

DOCUMENTS (1):
  • Informed Consent Form (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04417595/ICF_000.pdf